CLINICAL TRIAL: NCT04808934
Title: Stroke/Systemic Embolism and Major Bleeding in Patients Newly Treated With Oral Anticoagulants: a Real World Study From Portuguese Administrative Claims Data
Brief Title: NOAC Portuguese Real World Study
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn due to COVID19 pandemic. Several delays affected this study, therefore company decided to not conduct the study. It was cancelled prior to any enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001275
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Systemic Embolism; Major Bleeding
MeSH Terms: conditions — Stroke | interventions — apixaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Not applicable, this is a retrospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-Valvular Atrial Fibrillation (NVAF) Adults: Adult patients with NVAF newly treated with apixaban, dabigatran, rivaroxaban or VKAs between June 16, 2014 and December 31, 2018.
  Interventions: Drug: Apixaban; Drug: dabigatran; Drug: rivaroxaban; Drug: VKAs

INTERVENTIONS:
Drug: Apixaban — Adults receiving apixaban
Drug: dabigatran — Adults receiving dabigatran
Drug: rivaroxaban — Adults receiving rivaroxaban
Drug: VKAs — Adults receiving VKA

SUMMARY:
To determine if there is any difference in the effectiveness and safety outcomes of patients with NVAF newly treated with apixaban, dabigatran, rivaroxaban and vitamin K antagonists

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on the index date.
* At least 1 OAC (apixaban, dabigatran, rivaroxaban, VKAs) dispensed during the identification period.

Exclusion Criteria:

* Specialty of the physician responsible for the OAC prescription in the index date is one of the following: orthopedics, general surgery, vascular surgery or any other surgical specialty;
* Duration of OAC therapy during follow-up inferior to the cut-off defined during the feasibility assessment (except if the patient was admitted to in-hospital care during follow-up);
* The OAC dispensed in the index date was one of the following: dabigatran 75 mg or rivaroxaban 10 mg
* Hospital claims lacking a diagnosis code indicative of AF during the study period;
* Hospital claim indicating a diagnosis or procedure code indicative of pregnancy or childbirth during the study period;
* Hospital claim indicating a diagnosis or procedure code indicative of valvular heart disease, venous thromboembolism, cardiac surgery, pericarditis, hyperthyroidism and thyrotoxicity during the baseline period;
* Hospital claim indicating a diagnosis or procedure code indicative of hip and knee replacement surgery during the 6 weeks prior to the index date. Patients with past use of OAC will be excluded. Therefore, patients meeting any of the following criteria will be excluded:
* Had any OAC (apixaban, dabigatran, edoxaban, rivaroxaban, VKAs) dispensed during the 12-month baseline period;
* Had >1 OAC dispensed on the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients will be selected from the CCF database based on an apixaban, dabigatran, rivaroxaban or VKAs filled prescription between June 16, 2014 and December 31, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
stroke/systemic embolism event | between 2014 and 2018
  To compare the risk of stroke (either ischemic or hemorrhagic) or SE among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
major bleeding event | between 2014 and 2018
  To compare the risk of major bleeding (gastrointestinal [GI], intracranial [IC] and other) among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versusVKAs.

SECONDARY OUTCOMES:
ischemic stroke event | between 2014 and 2018
  To compare the risk of ischemic stroke among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
hemorrhagic stroke event | between 2014 and 2018
  To compare the risk of hemorrhagic stroke among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
systemic embolism event | 2014-2018
  To compare the risk of systemic embolism among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
major GI bleeding event | 2014-2018
  To compare the risk of major GI bleeding among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
major IC bleeding event | 2014-2018
  To compare the risk of major IC bleeding among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.
other major bleeding event | 2014-2018
  To compare the risk of other major bleeding among patients newly treated with each NOAC separately (apixaban, dabigatran, rivaroxaban) versus VKAs.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.